CLINICAL TRIAL: NCT04573647
Title: Evaluation of Changes in Corneal Stromal Thickness Using Anterior Segment OCT Following Treatment of Neurotrophic Ulcers With Oxervate
Brief Title: OCT Evaluation of Neurotrophic Ulcer Following Treatment With Oxervate
Status: Recruiting | Type: Observational
Sponsor: Sight Medical Doctors PLLC (Other)
Collaborators: Dompé, US, Inc. (Unknown)
Responsible Party: Principal Investigator, Brad Kligman, MD, Principle Investigator, Sight Medical Doctors PLLC
Other Study IDs: IIR-2019-1139
Record Dates: First submitted 2020-09-28; First posted 2020-10-05 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Neurotrophic Ulcer; Neurotrophic Keratitis; Neurotrophic Corneal Ulcer; Neurotrophic Keratoconjunctivitis
Keywords: Neurotrophic Ulcer; Neurotrophic Keratoconjunctivitis; Optical Coherence Tomography; OCT
MeSH Terms: interventions — cenegermin; Ophthalmic Solutions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Treatment group: All participants in this trial will be in the treatment group. They will administer Oxervate following the FDA approved guidelines: 1 drop to the affected eye 6 times per day for 8 weeks.
  Interventions: Drug: Cenegermin-Bkbj 0.002% Ophthalmic Solution [OXERVATE]

INTERVENTIONS:
Drug: Cenegermin-Bkbj 0.002% Ophthalmic Solution [OXERVATE] — Research subjects will use oxervate in affected eye following approved treatment regimen and have their eye measured with optical coherence tomography and a Cochet-Bonnet esthesiometer at various time points before, during and after treatment.

SUMMARY:
Neurotrophic keratitis (NK) is a condition where the cornea, or clear outer covering of the eye, has reduced sensation due to a variety of reasons. In more advanced cases of NK, the cornea can develop an area of thinning called an ulcer. The purpose of this research is to find out if Oxervate (cenegermin-bkbj 0.002%) an FDA-approved treatment for neurotrophic corneal ulcers leads to an increase in thickness of the corneal stroma (middle layer of the cornea) during and after treatment of a neurotrophic ulcer. Corneal thickness will be measured using optical coherence tomography (OCT), a non-contact imaging device used routinely in ophthalmology examinations. Corneal sensation will also be measured during and after treatment with a device called a Cochet-Bonnet esthesiometer to see if the treatment increases corneal sensation.

DETAILED DESCRIPTION:
Neurotrophic keratitis (NK) is a condition where the cornea, or clear outer covering of the eye, has reduced sensation due to a variety of reasons such as previous surgery or infection. In more advanced cases of NK, the cornea can develop an area of thinning called an ulcer. If the cornea becomes too thin, it is at risk for perforation or rupture, which requires extensive surgery to save vision and the eye. This risk can last for many years even after the ulcer is no longer active. The purpose of this research is to find out if Oxervate (cenegermin-bkbj 0.002%) an FDA-approved treatment for neurotrophic corneal ulcers leads to an increase in thickness of the corneal stroma (middle layer of the cornea) during and after treatment of a neurotrophic ulcer. The FDA trials demonstrated that Oxervate does lead to more rapid healing of the epithelium (thin surface layer) of the cornea, but it is unclear if it increases the thickness of the stroma, which is the strongest part of the cornea. Corneal thickness will be measured using optical coherence tomography (OCT), a non-contact imaging device used routinely in ophthalmology examinations. Corneal sensation will also be measured during and after treatment with a device called a Cochet-Bonnet esthesiometer to see if the treatment increases corneal sensation. If treatment with Oxervate increases corneal sensation, then this decreases the risk of future ulcer formation.

About 10 subjects will take part in this research.

ELIGIBILITY:
Inclusion Criteria:

* Neurotrophic keratitis with stage 3 neurotrophic ulcer (stromal thinning)
* Decreased corneal sensation relative to fellow eye determined qualitatively using wisp of cotton-tipped applicator to compare sensation in each eye without anesthesia.

Exclusion Criteria:

* Impending corneal perforation (descemetocele)
* Unable to physically complete diagnostic testing (cannot position head into slit lamp or OCT)
* Unable to commit to 6 month follow up prior to initiating study
* Unable to self-administer study drug following explanation and demonstration by PI and study coordinator
* Active infectious infiltrate clinically worsening by history or clinical appearance
* Pregnancy; patients must agree to use an acceptable form of birth control during study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults with stage 3 neurotrophic keratitis (ulcer)
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Stromal Thickness | 6 Months
  To determine with optical coherence tomography if stromal thickness at the thinnest point of a neurotrophic ulcer increases during and after treatment with Oxervate independent of corneal epithelium.

SECONDARY OUTCOMES:
Esthesiometry | 6 Months
  To quantitatively measure change in corneal esthesiometry during and after treatment of neurotrophic ulcers with Oxervate using Cochet-Bonnet esthesiometry
Clinical resolution of epithelial defects | 6 Months
  To evaluate time course of clinical resolution of epithelial defects in neurotrophic ulcers subjectively determined by slit lamp examination

CONTACTS AND LOCATIONS:
Overall Officials: Brad Kligman, MD, Principal Investigator — Sight Medical Doctors PLLC
Locations (1):
- SightMD, Manhasset, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sheha H, Tighe S, Hashem O, Hayashida Y. Update On Cenegermin Eye Drops In The Treatment Of Neurotrophic Keratitis. Clin Ophthalmol. 2019 Oct 7;13:1973-1980. doi: 10.2147/OPTH.S185184. eCollection 2019. PMID 31631965
- [Background] Micera A, Lambiase A, Puxeddu I, Aloe L, Stampachiacchiere B, Levi-Schaffer F, Bonini S, Bonini S. Nerve growth factor effect on human primary fibroblastic-keratocytes: possible mechanism during corneal healing. Exp Eye Res. 2006 Oct;83(4):747-57. doi: 10.1016/j.exer.2006.03.010. Epub 2006 May 23. PMID 16716299